CLINICAL TRIAL: NCT05633407
Title: A Phase 2 Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Efficacy and Safety of Efgartigimod IV in Adult Patients With Post-COVID-19 Postural Orthostatic Tachycardia Syndrome (POTS)
Brief Title: Efficacy and Safety Study of Efgartigimod in Adults With Post-COVID-19 POTS
Acronym: POTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARGX-113-2104
Record Dates: First submitted 2022-11-08; First posted 2022-12-01 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: POTS; Long COVID; Postural Orthostatic Tachycardia Syndrome; efgartigimod
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Post-Acute COVID-19 Syndrome | interventions — efgartigimod alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigimod (Experimental): Receive efgartigimod IV 10mg/kg during weekly infusions during a treatment period of 24 weeks
  Interventions: Drug: Efgartigimod
- Placebo (Placebo Comparator): Receive a matching placebo during weekly infusions during a treatment period of 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efgartigimod — Efgartigimod IV 10 mg/kg infusion qw for 24 weeks. Participants will be randomized to receive efgartigimod IV 10 mg/kg or matching placebo in a 2:1 ratio, respectively
  Arms: Efgartigimod
Drug: Placebo — Receive a matching placebo during weekly infusions during a treatment period of 24 weeks.
  Participants will be randomized to receive efgartigimod IV 10 mg/kg or matching placebo in a 2:1 ratio, respectively
  Arms: Placebo

SUMMARY:
The study aims to investigate the safety, tolerability, efficacy, pharmacodynamics (PD), pharmacokinetics (PK), and immunogenicity of efgartigimod compared to placebo in participants with post-COVID-19 postural orthostatic tachycardia syndrome (POTS) (post-COVID-19 POTS).

DETAILED DESCRIPTION:
The study aims to investigate the safety, tolerability, efficacy, pharmacodynamics (PD), pharmacokinetics (PK), and immunogenicity of efgartigimod compared to placebo in participants with post-COVID-19 postural orthostatic tachycardia syndrome (POTS) (post-COVID-19 POTS). Efgartigimod may be a viable treatment option for individuals diagnosed with post-COVID-19 POTS because it has been shown to reduce IgG levels, including IgG autoantibodies, which may underlie some of the autonomic disease manifestations in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Reached the age of consent when signing the informed consent form
2. Capable of providing signed informed consent and complying with protocol requirements
3. Diagnosed with new-onset POTS post-COVID-19 established by the following:

   1. History of COVID-19 based on a previous positive test result from either laboratory-confirmed COVID-19 test (eg, a PCR test) or non-laboratory-confirmed COVID-19 test (eg, rapid antigen test); this positive result may be either documented or patient-reported
   2. Tilt table or orthostatic vital sign measurements during screening consistent with consensus criteria: sustained HR increase of ≥30 bpm within 10 min of standing or head up tilt (≥40 bpm for individuals aged 18 to 19 years) and/or HR reaching >120 bpm within 10 min; absence of sustained 20 mmHg decrease in systolic blood pressure (SBP)
   3. Ongoing symptoms of POTS confirmed by the investigator with at least 3 symptoms in each of the following areas lasting longer than 12 weeks after either diagnosis of COVID-19 or after hospital discharge for COVID-19:

   i. Vasomotor symptoms: fatigue, orthostatic intolerance, brain fog, exertional dyspnea, difficulty with concentration, venous pooling, and exercise intolerance ii. Sympathetic over-compensation symptoms: palpitation, heat intolerance, nausea with or without vomiting, insomnia, anxiety, lack of appetite, chest pain, and diaphoresis
4. COMPASS 31 ≥35 at screening
5. Agree to use contraceptives consistent with local regulations regarding the methods of contraception for those participating in clinical studies and the following:

   Male participants: No male contraception is required Female participants of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline before receiving IMP. Contraceptive requirements.
6. Body mass index (BMI) <35 kg/m2

Exclusion Criteria:

1. Diagnosis of or receiving treatment for the following conditions before COVID-19: peripheral neuropathy, POTS, myalgic encephalomyelitis encephalitis/chronic fatigue syndrome, Ehlers Danlos syndrome confirmed by genetic testing, autonomic neuropathy, multiple sclerosis, stroke, spinal cord injury, or any known lesions in the central nervous system by imaging or neurological exam
2. History of or currently being treated for clinically significant ongoing cardiac arrythmia, heart failure, myocarditis, pulmonary embolism requiring anticoagulation, pulmonary fibrosis, or critical illness-related polyneuropathy or myopathy
3. Known autoimmune disease that, in the investigator's judgment, would interfere with an accurate assessment of clinical symptoms of post-COVID-19 POTS or puts the participant at undue risk
4. Known HIV disease or common variable immunodeficiency
5. History of malignancy unless considered cured by adequate treatment with no evidence of recurrence for ≥3 years before the first administration of IMP. Adequately-treated participants with the following cancers may be included at any time:

   1. Basal cell or squamous cell skin cancer
   2. Carcinoma in situ of the cervix
   3. Carcinoma in situ of the breast
   4. Incidental histological finding of prostate cancer (TNM stage T1a or T1b)
6. Clinically significant uncontrolled active or chronic bacterial, viral, or fungal infection or positive SARS-CoV-2 PCR test at screening
7. Positive serum test at screening for an active infection with any of the following:

   1. Hepatitis B virus (HBV) that is indicative of an acute or chronic infection, unless associated with a negative HB surface antigen (HBsAg) or negative HBV DNA test
   2. Hepatitis C virus (HCV) based on HCV antibody assay unless a negative RNA test is available
   3. HIV
8. A medical condition that could confound the results of the study or put the participant at undue risk in the investigator's judgment
9. Clinically significant disease, recent major surgery (within 3 months of screening), or intends to have surgery during the study; or any other condition that in the opinion of the investigator could confound the results of the study or put the participant at undue risk
10. Total IgG <4 g/L at screening
11. Received within 12 weeks or 5 half-lives (whichever is longer) before screening an investigational product
12. Received within 12 weeks before screening either intravenous immunoglobulin (Ig) IV or SC or plasmapheresis/plasma exchange (PLEX)
13. Received a live or live-attenuated vaccine less than 4 weeks before screening
14. Known hypersensitivity to IMP or 1 of its excipients
15. Previously participated in an efgartigimod clinical study and received at least 1 dose of IMP
16. Currently participating in another interventional clinical study
17. History (within 12 months of screening) of or current alcohol, drug, or medication abuse
18. Pregnant or lactating or intends to become pregnant during the study
19. Unwilling to remain on a stable regimen of medications during the study
20. Unwilling to avoid initiation of new physical rehabilitation or other physician-prescribed exercise programs during the 24-week treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of California, San Diego Sulpizio Cardiovascular Center, La Jolla, California
  - Stanford Movement Disorder Center, Palo Alto, California
  - Northshore University Health System, Glenview, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Harvard Medical School, Brigham and Women's Hospital, Boston, Massachusetts
  - Case Western Reserve University, Cleveland, Ohio
  - Vandetbilt University Medical Center / Clinical Research Center, Nashville, Tennessee
  - Apex Trials Croup, LLC, Fort Worth, Texas
  - Texas Institute of Cardiology, McKinney, Texas
  - Pioneer Clinical Research, Rosharon, Texas
  - Metrodora Institute, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dani M, Fedorowski A. Tackling POTS Needs More Than Just a Sympathetic Approach. Hypertension. 2024 Nov;81(11):2248-2250. doi: 10.1161/HYPERTENSIONAHA.124.23716. Epub 2024 Oct 16. No abstract available. PMID 39413203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase 2, randomized, double-blind study was conducted at 11 sites in the United States from 23-Sep-22 to 18-Apr-24 in participants with post-coronavirus disease 2019 (COVID-19) postural orthostatic tachycardia syndrome (POTS).
Pre-assignment Details: The study consisted of a screening period (approximately 4 weeks), a treatment period (24 weeks) and a follow-up period (approximately 8 weeks for participants who did not roll over to the open label extension study ARGX-113-2105 [NCT05918978). A total of 53 participants were randomized in a 2:1 ratio to receive either efgartigimod or matching placebo, respectively.
Groups:
- Efgartigimod: Participants received efgartigimod 10 milligram/kilogram (mg/kg) via intravenous (IV) infusion once weekly from Day 1 up to 24 weeks.
- Placebo: Participants received placebo matched to efgartigimod via IV infusion once weekly from Day 1 up to 24 weeks.
Period: Overall Study
Arm/Group | Efgartigimod | Placebo
Started | 36 | 17
Completed | 31 | 16
Not Completed | 5 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on full analysis set (FAS) which included all randomized participants who received at least 1 dose of study drug.
Groups:
- Efgartigimod: Participants received efgartigimod 10 mg/kg via IV infusion once weekly from Day 1 up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Efgartigimod | Placebo | Total
Number analyzed (Participants) | 36 | 17 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (12.82) | 36.8 (11.99) | 37.9 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 15 | 45
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 33 | 13 | 46
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 33 | 17 | 50
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in the COMPASS 31 (2-week Recall Version)
Description: Composite Autonomic Symptom Score (COMPASS) 31 modified version (2-week recall) is a self-rated questionnaire to evaluate the severity and distribution of autonomic symptoms in various autonomic nerve disorders. It consists of 31 questions in 6 weighted domains (orthostatic intolerance, vasomotor, secretomotor, gastrointestinal {GI}-mixed upper and diarrhea, bladder, and pupillomotor). A weighted total score of 0 (mild) to 100 (severe) was determined by adding a maximum raw score for each domain. Higher scores indicated a more severe degree of autonomic symptoms.
Time Frame: Baseline (Day 1) and Week 24
Population: The FAS included all randomized participants who received at least 1 dose of study drug. Only those participants with data collected at Baseline and Week 24 are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 22 | 15
score on a scale | -14.369 (15.2541) | -15.957 (17.2963)

2. Primary Outcome: Change From Baseline to Week 24 in the MaPS
Description: The Malmö POTS Symptom Score (MaPS) score is a dedicated POTS symptom scoring questionnaire. The score consists of 12 questions that assess symptom burden related (tachycardia, palpitations, dizziness, presyncope) and unrelated to orthostatic intolerance (GI symptoms, insomnia, concentration difficulties). Participants graded their symptoms for the past 7 days using a visual analog scale ranging from 0 (no symptoms) to 10 (worst possible). The total score was calculated by summing up the items/individual items and range was 0 to 120 points, with higher scores indicating more severe symptoms.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 22 | 15
score on a scale | -23.5 (25.87) | -19.8 (27.75)

3. Primary Outcome: Number of Participants With TEAEs and TESAEs
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. A serious adverse event (SAE) was any untoward medical occurrence that at any dose resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or any other medically important event. Treatment-emergent adverse events (TEAEs) were defined as AEs with onset on or after the first administration of study drug up to and including 60 days after the last study drug administration.
Time Frame: From the first dose of study drug (Day 1) up to 60 days post last dose of study drug, up to 236 days
Population: The safety analysis set (SAF) included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 36 | 17
Participants
  TEAEs | 31 | 14
  TESAEs | 0 | 0

4. Secondary Outcome: Percentage of Participants With Improved PGI-S at Week 24
Description: The Patient Global Impression-Severity (PGI-S) is a participant-rated, single-item scale to assess the severity of a health condition. The scale was used to assess the severity of symptoms over the past week (1-week recall) and overall experience of symptoms over the past 2 weeks (2-week recall). Both were rated on a 4-point type Likert scale, with scores ranging from 1 (none), 2 (mild), 3 (moderate), and 4 (severe). Higher scores indicate greater symptom severity. An "improved PGI-S" was defined by a change from baseline of -3, -2 and -1.
Time Frame: Baseline (Day 1) and Week 24
Population: The FAS included all randomized participants who received at least 1 dose of study drug. Only participants with available data at week 24 are included.
Measure: Number; unit: percentage of participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 22 | 15
percentage of participants
  1-week recall | 45.5 | 53.3
  2-week recall | 54.5 | 33.3

5. Secondary Outcome: Percentage of Participants With Improved in PGI-C at Week 24
Description: The Patient Global Impression-Change (PGIC) is a single-item scale to capture the participant's perception of a change in their overall symptom severity. Overall change in symptoms was rated on a 7-point Likert scale, with scores ranging from 1 (much better), 2 (somewhat better), 3 (a little better), 4 (no change), 5 (a little worse), 6 (somewhat worse), and 7 (much worse). Higher PGI-C scores signify worse outcome. An "improved PGI-C" was defined by a change from baseline of 1, 2 and 3.
Time Frame: Baseline (Day 1) and Week 24
Population: The FAS included all randomized participants who received at least 1 dose of study drug. Only participants with data available for week 24 are included.
Measure: Number; unit: percentage of participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 26 | 15
percentage of participants | 65.4 | 53.3

6. Secondary Outcome: Change From Baseline to Week 24 in the PROMIS Fatigue Short Form 8a
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 8a assesses the impact and perceived fatigue during the last 7 days. This validated 8-question scale has 5 response options, with scores ranging from 1 (not at all) to 5 (very much). Total scores ranged from 8 to 40; higher scores indicated higher fatigue levels and were converted to a T-score with a mean of 50 and standard deviation of 10. A decrease in T-score (negative change from baseline) indicated improvement in fatigue.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 22 | 15
T-score | -9.5 (8.77) | -7.0 (9.40)

7. Secondary Outcome: Change From Baseline to Week 24 in the PROMIS Cognitive Function Short Form 6a
Description: PROMIS Cognitive Function Short Form 6a assesses the frequency of cognitive difficulties experienced in the past 7 days. The questionnaire comprises 6 questions on subjective cognitive difficulties regarding a participant's concentration, memory, language, mental acuity, and perceived changes in cognitive functioning. The participant marks their response on a 5-point Likert scale (1: never and 5: very often). Scores ranged from 6 to 30; higher scores indicated worse perceived cognitive functioning and were converted to a T-score with a mean of 50 and standard deviation of 10. An increase in T-score (positive change from baseline) indicated better cognitive function.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 22 | 15
T-score | 3.9 (9.58) | 6.7 (9.74)

8. Secondary Outcome: Percent Change From Baseline in Total IgG Levels at Week 24
Description: Blood samples for immunoglobulin G (IgG) analysis were collected at specified time points. Total IgG concentrations were quantified using validated methods at a central laboratory.
Time Frame: Baseline (Day 1) and Week 24
Population: The SAF included all randomized participants who received at least 1 dose of study drug. Only those participants with data collected at Baseline and Week 24 are reported.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 27 | 14
percent change | -69.341 (6.0637) | 5.868 (13.1379)

9. Secondary Outcome: Serum Concentration of Efgartigimod
Description: Serum samples were collected at specified timepoints to determine the concentration of efgartigimod.
Time Frame: Pre-dose and post-dose at Baseline (Day 1), Weeks 1, 4, 12 and at Week 24
Population: The pharmacokinetic (PK) analysis set included all randomized participants who received at least 1 dose of efgartigimod and had at least 1 measured concentration of efgartigimod at a scheduled PK time point after start of dosing without protocol violations or events with potential to affect the PK concentration. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanogram (ng)/mL
Arm/Group | Efgartigimod
Number analyzed (Participants) | 34
nanogram (ng)/mL
  Baseline, pre-dose | NA (NA) — NA indicates that the mean and standard deviation were below the lower limit of quantification (LLOQ). LLOQ was 200 ng/mL.
  Baseline, post-dose: number analyzed (Participants) | 28
  Baseline, post-dose | 260536 (235110)
  Week 1, pre-dose: number analyzed (Participants) | 30
  Week 1, pre-dose | 10711 (3580)
  Week 1, post-dose: number analyzed (Participants) | 26
  Week 1, post-dose | 235100 (68316)
  Week 4, pre-dose: number analyzed (Participants) | 33
  Week 4, pre-dose | 12612 (5631)
  Week 4, post-dose: number analyzed (Participants) | 26
  Week 4, post-dose | 230308 (54329)
  Week 12, pre-dose: number analyzed (Participants) | 28
  Week 12, pre-dose | 18966 (39993)
  Week 12, post-dose: number analyzed (Participants) | 25
  Week 12, post-dose | 216760 (56621)
  Week 24: number analyzed (Participants) | 25
  Week 24 | 10450 (3894)

10. Secondary Outcome: Number of Participants With ADAs Against Efgartigimod
Description: Blood samples were collected at specified timepoints to assess anti-drug antibodies (ADAs) against efgartigimod. ADA incidence reported here was defined as total number of participants with treatment-induced and treatment-boosted ADA. Treatment-induced ADA was defined as a baseline negative sample and at least 1 positive post-baseline sample. Treatment-boosted ADA was defined as a baseline positive sample and the titer value increased 4-fold or more compared to baseline.
Time Frame: Up to Week 24
Population: The SAF included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 36 | 17
Participants | 5 | 1

ADVERSE EVENTS:
Time Frame: From the first dose of study drug (Day 1) up to 60 days post last dose of study drug, up to 236 days.
Description: Analysis was performed on the SAF. Laboratory abnormalities were reported as AEs.
Arm/Group | Efgartigimod | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/17
Other Adverse Events (participants affected / at risk) | 31/36 | 14/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efgartigimod (N=36) | Placebo (N=17)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (4)
Mydriasis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (6) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (13) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (4) | 0 (0)
Fatigue (General disorders) | 10 (13) | 3 (7)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Infusion site bruising (General disorders) | 0 (0) | 2 (2)
Infusion site pain (General disorders) | 1 (1) | 2 (2)
Injection site oedema (General disorders) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Overgrowth bacterial (Infections and infestations) | 0 (0) | 1 (1)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (6) | 2 (3)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 2 (2) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 3 (5)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 10 (20) | 3 (6)
Migraine (Nervous system disorders) | 2 (2) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (4)
Neuralgia (Nervous system disorders) | 1 (6) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT05633407/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT05633407/SAP_001.pdf